CLINICAL TRIAL: NCT04061083
Title: Effects of Three Endotracheal Tube Cuff Pressure Control on Microaspiration of Gastric Contents: a Randomized Controlled Trial
Brief Title: Effects of Endotracheal Tube Cuff Pressure Control on Microaspiration of Gastric Contents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Afyonkarahisar Health Sciences University Hospital (Unknown)
Responsible Party: Principal Investigator, Özlem SOYER, Research Assisstant, Msc, RN, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 118S409
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Mechanical Ventilation Complication; Ventilator Associated Pneumonia; Nursing Caries; Aspiration, Respiratory
Keywords: Intensive Care
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous Endotracheal Cuff Pressure Control (Experimental): Continuous endotracheal cuff pressure control using smart cuff manager during the first 48 hours of intubation in the intensive care unit
  Interventions: Device: Smart Cuff Manager
- Intermittent Endotracheal Cuff Pressure Control (Experimental): Intermittent cuff pressure control through manual manometer measurement performed 3 times per day during the first 48 hours of intubation in the intensive care unit
  Interventions: Device: Manometer
- Standard Care (No Intervention): ET cuff pressure control will be provided with pilot balloon fingers during the first 48 hours of intubation in the intensive care unit

INTERVENTIONS:
Device: Smart Cuff Manager — Participant will be attached to the smart cuff manager within 4 hours after intubation. They will remain attached during the first 48 hours of intubation in the intensive care unit
  Arms: Continuous Endotracheal Cuff Pressure Control
Device: Manometer — Participant will be attached to the manometer within 4 hours after intubation. They will assess 3 times per day during the first 48 hours of intubation in the intensive care unit
  Arms: Intermittent Endotracheal Cuff Pressure Control

SUMMARY:
The purpose of study is to determine effects of three different ET cuff pressure control on microaspiration of the stomach contents.

DETAILED DESCRIPTION:
In the study, ET cuff pressure control will be provided with pilot balloon fingers (Control Group), intermittent with a manometer (Study Group 1) and continuously with a smart cuff manager (Study Group 2).

To assess the effect of different ETT cuff pressure control on microaspiration of the stomach contents, the pepsin level will be measured during deep tracheal secretions. The samples will be examined in the first four hours after intubation, all secretions collected up to the 24th hour of intubation after first sample intake and all secretions collected between 24-48 hours after intubation. Pepsin level will be considered as positive for cut-off point. In addition, the effect of different ETT cuff pressures control on the incidence of VAP will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering of the patient or relatives who will participate in the study,
* Patients who require mechanical ventilation support with endotracheal tube supply for 48 hours.

Exclusion Criteria:

* Patients who are contraindicated in giving a semi-fowler position,
* Patients with enteral nutrition contraindications,
* Patients connected to mechanical ventilators for more than 48 hours,
* Patients with tracheostomy,
* Patients admitted to ICU for gastroesophageal reflux disease, aspiration pneumonia or suspicion,
* Nasal endotracheal intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Microaspiration of Gastric Contents | From randomisation to 48 hours after intubation
  The unintentional aspiration of very small amounts of gastric contents

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem SOYER, Afyonkarahisar, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Er OS, Van Giersbergen MY, Celik S. Effects of three endotracheal tube cuff pressure control measures on microaspiration of gastric content: Study protocol for randomised controlled trial. J Clin Nurs. 2023 Apr;32(7-8):1476-1486. doi: 10.1111/jocn.16493. Epub 2022 Aug 24. PMID 36002981

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT04061083/Prot_SAP_000.pdf